CLINICAL TRIAL: NCT04121988
Title: Prospective Observational Study of Diagnostic Yield in Cushing's Disease Using Deep Learning Based Denoising MRI
Brief Title: Diagnostic Yield of Deep Learning Based Denoising MRI in Cushing's Disease
Status: Terminated | Type: Observational
Why Stopped: Patients recruitment was difficult and the primary author quitted her role.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Sung Kim, Professor, Asan Medical Center
Other Study IDs: AsanMCHSKim_04
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pituitary ACTH Secreting Adenoma
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Denoising MRI group: Patients suspected of Cushing disease undergoing deep learning based denoising MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — 1 mm slice thickness with deep learning based reconstruction algorithm applied to the following sequences:
  * Coronal T2 weighted imaging
  * Dynamic contrast enhanced T1 weighted imaging
  * Coronal contrast enhanced T1 weighted imaging

SUMMARY:
Negative MRI findings may occur in up to 40% of cases of ACTH producing microadenomas. The aim of the study is to evaluate if detection of ACTH producing microadenomas can be increased using deep learning based denoising MRI.

DETAILED DESCRIPTION:
Detecting ACTH producing microadenoma in MRI is important in establishing the diagnosis of Cushing disease and may enable patients to avoid additional diagnostic tests such as inferior petrosal sinus sampling. However, detecting ACTH producing microadenoma in MRI remains as a diagnostic challenge due its small size with its median diameter of 5-mm. Many attempts have been made in order to improve the sensitivity of detecting ACTH producing microadenoma. It is generally accepted as standard clinical practice to perform dynamic contrast enhanced T1 weighted image to delineate delayed enhancing microadenonoma in comparison to the background enhancement of the normal gland. Despite these attempts, negative MRI findings may occur in up to 40% of cases of ACTH producing microadenomas and there is a need to improve its detection rate. Theoretically, performing thin slice thickness scans should help detecting the lesion but this is unavoidably accompanied with increased level of noise. Deep learning based denoising algorithm can be applied to reduce the noise level and potentially increase the detection rate of ACTH producing microadenomas. The aim of the study is to evaluate if detection of ACTH producing microadenomas can be increased using deep learning based denoising MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of Cushing disease undergoing MRI
* Signed informed consent

Exclusion Criteria:

* Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulates, electronic infusion pumps, etc), because such devices may be displaced or malfunction
* Patients who are pregnant or breast feeding; urine pregnancy test will be performed on women of child bearing potential
* Poor MRI image quality due to artifacts

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of tertiary hospital center
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Detection rate of ACTH producing microadenoma | 2 months
  Proportion of positive MRI with visible microadenoma as percentage (%)

SECONDARY OUTCOMES:
Proportion of patients undergoing additional diagnostic tests | 6 months
  Proportion of patients undergoing additional diagnostic tests as percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sung Kim, MD PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grober Y, Grober H, Wintermark M, Jane JA, Oldfield EH. Comparison of MRI techniques for detecting microadenomas in Cushing's disease. J Neurosurg. 2018 Apr;128(4):1051-1057. doi: 10.3171/2017.3.JNS163122. Epub 2017 Apr 28. PMID 28452619
- [Background] Law M, Wang R, Liu CJ, Shiroishi MS, Carmichael JD, Mack WJ, Weiss M, Wang DJJ, Toga AW, Zada G. Value of pituitary gland MRI at 7 T in Cushing's disease and relationship to inferior petrosal sinus sampling: case report. J Neurosurg. 2018 Mar 23;130(2):347-351. doi: 10.3171/2017.9.JNS171969. Print 2019 Feb 1. PMID 29570013